CLINICAL TRIAL: NCT00291460
Title: Randomized Controlled Trial of Inspiratory Muscle Training in Patients With Stable Hypercapnic Respiratory Failure Due to COPD
Brief Title: Inspiratory Muscle Training in Hypercapnic COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krankenhaus Kloster Grafschaft (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FKKG IMT 0106
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2006-02

CONDITIONS: COPD; Respiratory Failure
Keywords: COPD; respiratory failure; inspiratory muscle training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

INTERVENTIONS:
Device: inspiratory muscle training

SUMMARY:
The trial intends to investigate, whether inspiratory muscle training in hypercapnic patients improves inspiratory muscle strength, inspiratory muscle endurance and endurance to walk within six minutes.

DETAILED DESCRIPTION:
Inspiratory muscle training is known to improve inspiratory muscle strength, inspiratory muscle endurance and walking distance within six minutes in patients with neuromuscular and thoraco-restrictive disease as well as in patients with COPD. Studies have only been conducted in patients without established respiratory failure. COPD patients with respiratory failure though are characterized by higher work rates of the inspiratory muscles and higher esophageal pressure swings compared to non-hypercapnic patients indication a discrepancy between muscle load and muscle capabilities. Therefore we hypothesize that for these patients training of their inspiratory muscles will be of benefit in terms of improvement of muscular and whole body endurance.

During this investigation inspiratory muscle training will be applied in a randomized controlled fashion in 40 patients over a period of four weeks parallel to physical rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* COPD with FEV1/FVC < 70 %
* age > 18
* stable disease
* able to walk
* carbon dioxide >= 48 mmHg

Exclusion Criteria:

* ejection fraction of the heart < 40 %
* active psychiatric disease
* bronchial hyperresponsiveness according to ATS criteria
* pregnancy
* renal insufficiency with a creatinine < 2 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-02; Study Completion 2008-03

PRIMARY OUTCOMES:
inspiratory muscle strength
inspiratory muscle endurance
walking distance with dyspnea score
Carbon dioxide level

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dellweg, M.D., Principal Investigator — FKKG; Dieter Koehler, Prof. Dr., Study Chair — FKKG
Locations (1):
- Fachkrankenhaus Kloster Grafschaft, Schmallenberg, Germany